CLINICAL TRIAL: NCT04485780
Title: The Optimal Timing of Botulinum Toxin Injection for Pain Control in Patients Undergoing Hemorrhoidectomy-A Prospective, Randomized Study
Brief Title: Botulinum Toxin Injection in Patients Undergoing Hemorrhoidectomy-A Prospective, Randomized Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yi-Chiao Cheng, Attending surgeon, division of colon and rectal surgery, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1-107-05-042
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: The Influence of Timing of Botulinum Toxin Injection on Postoperative Pain Control
Keywords: hemorrhoidectomy; botulinum toxin; pain; wound healing
MeSH Terms: conditions — Pain | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulinum toxin injection during surgery (Placebo Comparator): Patients in this group underwent Botulinum toxin injection during surgery
  Interventions: Biological: botulinum toxin type A
- Botulinum toxin injection one week before surgery (Experimental): Patients in this group underwent Botulinum toxin injection at the outpatient clinic one week before surgery
  Interventions: Biological: botulinum toxin type A

INTERVENTIONS:
Biological: botulinum toxin type A — In the outpatient department, patients who need hemorrhoidectomy were randomly assigned to two groups at a 1:1 ratio using a computer-generated list of random numbers (Microsoft Excel). One group received Botulinum toxin injection during the outpatient clinic one week before the operation(experimental group, EG), and the other group received injection during the operation(control group, CG). The two groups were compared for the influence of postoperative pain control and wound healing rate.
  Other Names: Botox

SUMMARY:
This is a prospective, randomized study, which anticipatedly recruited 60 patients in the outpatient department who need hemorrhoidectomy from January 2019 to December 2019. After obtaining those patients' consent in the clinic, they were randomly assigned to two groups at a 1:1 ratio using a computer-generated list of random numbers (Microsoft Excel). One group received Botulinum toxin injection during the outpatient clinic one week before the operation(experimental group, EG), and the other group received injection during the operation(control group, CG). The two groups were compared for the influence of postoperative pain control and wound healing rate.

ELIGIBILITY:
Inclusion Criteria:

* patients with age over 20 but under 80, who need to undergo hemorrhoidectomy

Exclusion Criteria:

* patients under the age of 20
* patients with nonsteroidal anti-inflammatory drugs (NSAIDs) allergy or sensitivity
* patients with Botulinum toxin allergy or sensitivity
* patients with dialysis or renal insufficiency
* pregnant and breastfeeding women
* vulnerable population

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-10-08 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
one week after operation | 1 weel
  The degree of postoperative pain is assessed by visual analog scale (VAS). After operation, we record patients' average VAS score and maximum VAS score every day until one week after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, National Defense Medical Center, Taipei, Taiwan

REFERENCES:
- [Derived] Cheng YC, Beh JY, Wu PH, Tsai NY, Jao SW. Early botulinum toxin injection reduces pain after hemorrhoidectomy: a pilot study. Tech Coloproctol. 2022 Jan;26(1):53-60. doi: 10.1007/s10151-021-02542-4. Epub 2021 Oct 27. PMID 34705137